CLINICAL TRIAL: NCT05185219
Title: The Effect of Valerian on Insomnia in Menopausal Women: Randomized Placebo-controlled Trial
Brief Title: The Effect of Valerian on Insomnia in Menopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shan-Yu Su, Director, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021MenoVal / CMUH109-REC2-177
Record Dates: First submitted 2021-12-03; First posted 2022-01-11 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Menopausal Women; Insomnia
Keywords: menopause; insomnia; valerian
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valerian (Experimental): generic name: XIE CAO CONC dosage form: capsule dosage: 500 mg/capsule, 6 capsules a day frequency: 3 times a day after each meal, 2 capsules each time duration: 30 days
  Interventions: Drug: Valerian
- Control (Placebo Comparator): generic name: placebo (Caramel Colors dyed starch) dosage form: capsule dosage: 500 mg/capsule, 6 capsules a day frequency: 3 times a day after each meal, 2 capsules each time duration: 30 days
  Interventions: Drug: Valerian

INTERVENTIONS:
Drug: Valerian — A natural plant

SUMMARY:
Menopausal women often complain that it is difficult to fall asleep and easy to wake up at night and early in the morning and it is in the middle of night difficult to fall asleep again. If the above symptoms persist for at least three months and occur at least three times a week, plus the impact on daytime work and rest, and meet the International Classification of Sleep Disorders (ICSD-3) )'S s "Insomnia" diagnostic criteria. According to statistics, 30% to 60% of women face sleep disorders during menopause.

DETAILED DESCRIPTION:
The investigators expect to receive outpatient admissions in the hospital attached to China Medical University. Menopausal women aged 45-60 years old who have been diagnosed with insomnia who meet criteria of International Classification of Sleep Disorders (ICSD-3) will be randomly assigned for clinical trials. Patients will take two Valerian capsules (1000mg/day) per day for four weeks. Pittsburgh Sleep Index (PSQI) will be used to evaluate subjective sleep quality. TCM patterns will be evaluated by three physicians of TCM gynecology independently before and after taking Valeriana. The data will conduct a biological analysis to compare the difference in sleep quality between the trial group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. 45〜60 years old, and is menopaused for at least 1 year。
2. meet the criteria of ICSD-3 for insomnia
3. PSQI > 5

Exclusion Criteria:

1. psychiatry disease
2. Heart, brain, liver diseases
3. Insomnia is caused by diseases.
4. Steroid used within 6 months
5. pregnant or breastfeeding

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female-specific condition
Enrollment: 100 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Sleep quallity | 30 days
  Sleep quality will be evaluated by Pittsburgh Sleep Index (PSQI). The sum of the scores on PSQI ranges from 0 to 21, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Traditional Chinese medicine (TCM) constitution | 30 days
  TCM constitution will be measured by three TCM doctor and TCM questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No